CLINICAL TRIAL: NCT01953744
Title: Phase 3 Randomized Trial Comparing Fluconazole to Meglumine Antimoniate in the Treatment of Cutaneous Leishmaniasis Caused by L. Braziliensis and L. Guyanensis
Brief Title: High Dose Fluconazole in Cutaneous Leishmaniasis in Bahia and Manaus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low cure rate in the study (fluconazole) group
Sponsor: Hospital Universitário Professor Edgard Santos (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Federal University of Bahia (Other)
Responsible Party: Principal Investigator, Paulo Roberto Lima Machado, Associate Researcher, Hospital Universitário Professor Edgard Santos
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FlucoLBrBaMa
Record Dates: First submitted 2013-09-25; First posted 2013-10-01 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Cutaneous Leishmaniasis
Keywords: Fluconazole; Meglumine antimoniate;L.Braziliensis;; L.Guyanensis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Fluconazole; Meglumine Antimoniate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluconazole (Experimental): Fluconazole will be administered by oral route at 6-8mg/kg/day during 28 days.
  Interventions: Drug: Fluconazole
- Meglumine Antimoniate (Active Comparator): Meglumine Antimoniate will be administered by intravenous route at 20mg/kg/day during 20 days.
  Interventions: Drug: Meglumine Antimoniate

INTERVENTIONS:
Drug: Fluconazole — Fluconazole is presented in 150mg capsules and will be administered by oral route at a dosage of 6-8mg/kg/day during 28 days.
  Arms: Fluconazole
Drug: Meglumine Antimoniate — Meglumine Antimoniate will be administered as the standard treatment for cutaneous leishmaniasis by intravenous route at a dosage of 20mg/kg/day, during 20 days.
  Other Names: Glucantime
  Arms: Meglumine Antimoniate

SUMMARY:
The purpose of this study is to evaluate the therapeutic response to fluconazole in patients with cutaneous leishmaniasis caused by and L.(V.)guyanensis and L.(V.) braziliensis.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed (untreated) cutaneous leishmaniasis with localized lesions and a positive culture or diagnosed by polymerase chain reaction (PCR) methods or by intradermal skin testing (Montenegro test).
* Number of lesions: 1 to 3 ulcerative lesions.
* Lesion´s diameter: 1 to 5 cm.
* Disease duration: up to three months.

Exclusion Criteria:

* Evidence of serious underlying disease (cardiac, renal, hepatic or pulmonary)
* Immunodeficiency or antibody to HIV
* Any non-compensated or uncontrolled condition, such as active tuberculosis, malignant disease, severe malaria, HIV, or other major infectious diseases
* Lactation, pregnancy (to be determined by adequate test) or inadequate contraception in females of childbearing potential for treatment period plus 2 months

  * Lack of suitability for the trial:
* Negative parasitology (aspirate/biopsy/PCR)or negative Montenegro test
* Any history of prior anti-leishmania therapy
* Any condition which compromises ability to comply with the study procedures

  * Administrative reasons:
* Lack of ability or willingness to give informed consent (patient and/or parent / legal representative)
* Anticipated non-availability for study visits/procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2014-02; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Cure rate or complete cicatrization of the ulcer. | 6 months
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients.

SECONDARY OUTCOMES:
Initial cure rate or complete cicatrization of the ulcer | 2 months
  All lesions will be categorized as either active or healed (cured) at follow-up visits. Only lesions with complete re-epithelialization, without raised borders, infiltrations or crusts will be considered healed. Evaluation of the lesions will be performed by 2 clinicians who will be unaware of the group assignment of all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Roberto Lima Machado, PhD, Principal Investigator — University of Bahia
Locations (1):
- Posto de Saúde de Corte de Pedra, Presidente Tancredo Neves, Estado de Bahia, Brazil

REFERENCES:
- [Derived] Prates FV, Dourado ME, Silva SC, Schriefer A, Guimaraes LH, Brito MD, Almeida J, Carvalho EM, Machado PR. Fluconazole in the Treatment of Cutaneous Leishmaniasis Caused by Leishmania braziliensis: A Randomized Controlled Trial. Clin Infect Dis. 2017 Jan 1;64(1):67-71. doi: 10.1093/cid/ciw662. Epub 2016 Nov 1. PMID 27803094